CLINICAL TRIAL: NCT04081428
Title: Using Breath,Cell Free DNA and Image Analysis to PRedIct Normal TissUe and Tumour Response During Prostate Cancer SBRT With RayPilot® Motion Management
Brief Title: Using Breath, Cell Free DNA and Image Analysis to PRedIct Normal TissUe and Tumour Response During Prostate Cancer SBRT
Acronym: PRINToUT
Status: Active, not recruiting | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC18048
Record Dates: First submitted 2019-08-01; First posted 2019-09-09 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer; Radiotherapy Side Effects; Volatile Organic Compounds; DNA Damage
Keywords: Prostate cancer; Cell free DNA; Volatile organic compounds; Stereotactic Body Radiotherapy; Radiotherapy side effects; Imaging biomarkers
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery; Cell-Free Nucleic Acids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Volatile Organic Compound Breath Analysis, Cell-Free DNA normal tissue and tumour DNA, Cone Beam CT pre and post each fraction of radiotherapy, Genomic saliva analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — Daily collection of breath and blood before and after each of the 5 radiotherapy treatment sessions. Before and after daily cone beam CT image collection
  Other Names: Breath Analysis; Cell-free DNA; Imaging biomarkers; Treatment image guidance with the RayPilot®

SUMMARY:
Personalisation of radiotherapy dose based on real-time assessments of normal tissue and tumour response would maximise cure and minimise treatment related toxicity. During a 5 fraction course of prostate Stereotactic Body Radiotherapy (SBRT) this pilot study will assess whether a number of different biomarker approaches can predict for normal tissue and tumour response. Firstly the investigators will analyse volatile organic compounds released within the breath with each fraction of treatment. Secondly the investigators will analyse cell free normal tissue and tumour DNA released during treatment. Thirdly the investigators will develop imaging processing algorithms to look for imaging biomarkers predicting rectal wall toxicity using pre and post treatment cone beam CT verification images. Each of these approaches will be assessed against prostate specific antigen (PSA), Common Terminology Criteria for Adverse Events (CTCAE v4.0) criteria and Expanded Prostate Cancer Index Composite (EPIC-26) patient reported outcomes with a maximum of 24 months of follow up.

DETAILED DESCRIPTION:
Radiotherapy scheduling and prescription dose does not take into account individual patient heterogeneity in normal tissue response or tumour response. Personalisation of radiotherapy dose based on real-time assessments of normal tissue and tumour response would maximise cure and minimise treatment related toxicity. During a 5 fraction course of prostate Stereotactic Body Radiotherapy (SBRT) this pilot study will assess whether a number of different biomarker approaches can predict for normal tissue and tumour response. Firstly the investigators will analyse volatile organic compounds released within the breath with each fraction of treatment using Gas Chromatography Ion Mobility Spectroscopy (GC-IMS). The investigators have extensive experience in this area within the TOXI-Triage research program (www.toxi-triage.eu/) including deep learning and machine learning techniques to interrogate the metabolomics data generated. Secondly the investigators will analyse cell free normal tissue and tumour DNA released during treatment to assess both tumour and normal tissue response. Radiotherapy releases large amounts in to the blood stream allowing easier quantitative analysis. Thirdly the investigators will look for imaging biomarkers of rectal wall toxicity using imaging analysis algorithms of on-treatment cone beam verification CT images taken before and after each radiotherapy treatment. The RayPilot® system made by Micropos Medical Ltd tracks prostate motion throughout the SBRT delivery to ensure that the treatment dose is delivered with great precision. The potential of each biomarker approach for predicting normal tissue and tumour response will be assessed against PSA and CTCAE v 4.0 toxicity criteria and EPIC-26 patient reported outcome measures after 24 months of patient follow up.

ELIGIBILITY:
Inclusion Criteria:

* Low risk prostate cancer T1-2, PSA<10ng/ml, Gleason score (GS) 3+3=6
* Intermediate risk prostate cancer T1-T2, PSA 10-20ng/ml,GS ≤7(3+4=7 only)
* World Health Organisation (WHO) performance status 0-2
* Prostate volume ≤90cc
* International Prostate Symptom Score (IPSS) ≤20
* Peak urinary flow rate (Q-max) >10cc/sec
* Urinary residual <250mls total
* No prior Trans Urethral Resection of the Prostate (TURP)
* No previous pelvic radiotherapy
* Able to give informed consent
* Aged between 18-85 years of age

Exclusion Criteria:

* Inflammatory bowel disease
* Previous androgen deprivation therapy
* History of urinary retention

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — men with prostate cancer
Study Population: Men diagnosed with localised prostate cancer within the South East of Scotland cancer network who are suitable for study entry
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2026-01-11 (Estimated); Study Completion 2026-01-11 (Estimated)

PRIMARY OUTCOMES:
Measurement of the relative change in Gas Chromatography Ion Mobility Spectra (GC-IMS) of Volatile Organic Compounds (VOC's) from breath samples of men with prostate cancer treated with prostate stereotactic body radiotherapy (SBRT) | pre treatment before each fraction of SBRT day 1 to day 5, then at 1 and 3 hours post treatment day 1 to day 5
  Measurement of the change in the 3D chromatogram of volatile organic compound GC-IMS Spectra detected from baseline pre-treatment, to completion of SBRT at each time point, for each patient. Each 3D chromatogram GC-IMS printout is generated from the readings of each axis. The y axis is associated with GC separation of VOC's, the x axis measures the movement of the generated ions (IMS drift time) and the z axis ion detector response equating to concentration. These 3 values separate, identify and quantify the VOC compounds detected.
Measurement of the relative change in normal tissue and tumour cell free DNA (cfDNA) released into the blood of men with prostate cancer treated with prostate stereotactic body radiotherapy (SBRT) | pre treatment before each fraction of SBRT day 1 to day 5, then at 1 and 3 hours post treatment day 1 to day 5
  Change in the density of 90-150 base pair fragment size cfDNA from baseline pre-treatment to completion of SBRT for each time point, for each patient
Measurement of the true rectal wall delivered radiation dose compared to planned dose during the prostate SBRT for each patient | Immediately pre each fraction of SBRT day 1 to 5 and immediately post each fraction of SBRT day 1 to 5
  Dose calculation in cGy between expected and observed actual dose to the rectal wall using pre and post each fraction radiotherapy linear accelerator treatment verification cone beam CT scans

SECONDARY OUTCOMES:
Measurement of SBRT treatment related acute and late normal tissue toxicity | Baseline, completion of SBRT, week 6, then 3 months, 6 months, 12 months, 18 months and 24 months post treatment
  Common Terminology Criteria for Adverse Events CTCAE v 4.0 scores for urinary and bowel treatment related toxicity. Scale runs form Grade 1 mild requiring no intervention to grade 5 death
Measurement of SBRT treatment related quality of life | Baseline, completion of SBRT, week 6, then 3 months, 6 months, 12 months, 18 months and 24 months post treatment
  Expanded Prostate Cancer Index Composite EPIC-26 patient reported outcomes questionnaire. A clinical tool to assess urinary, bowel, sexual and vitality health. The score from each of the 5 domains runs from 0 (none) to 12 (severe) impact on quality of life. Each domain score when added together gives an overall score of zero (unaffected) to 60 (severely affected)

CONTACTS AND LOCATIONS:
Overall Officials: Duncan B McLaren, MBBS, Principal Investigator — NHS Lothian
Locations (1):
- Edinburgh Cancer Centre, Western General Hospital, Edinburgh, Mid Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The pilot data will be used to inform a larger study cohort and to establish the optimal methodology and time points for sample collection